CLINICAL TRIAL: NCT04280276
Title: Utilizing TruGraf Testing in Recipients of Kidney Transplantation With High Intra-patient Variability in Tacrolimus Exposure: A Pilot Study
Brief Title: TruGraf Utilization in High IPV Levels
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor, TGI, was acquired by Eurofins Inc. New owner requested all IIT's be terminated.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Transplant Genomics, Inc. (Industry)
Responsible Party: Principal Investigator, Roberto Kalil, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00089343
Record Dates: First submitted 2020-02-11; First posted 2020-02-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Patients with high IPV (designated as ≥ 30%). (Active Comparator): Patients with high IPV (designated as ≥ 30%).
  Interventions: Diagnostic Test: TruGraf test
- Group 2 - patients with normal IPV (< 30%). (Active Comparator): Patients with normal IPV (< 30%). Will assess risk of subclinical acute rejection in patients with high IPV compared to normal IPV. All tacrolimus 12 h trough levels in patients with stable allograft function at least 3 months post-transplant.
  Interventions: Diagnostic Test: TruGraf test

INTERVENTIONS:
Diagnostic Test: TruGraf test — To obtain longitudinal TruGraf testing in patients with stable creatinine, high and normal IPV in tacrolimus levels, between 3 and 18 months post-transplant at the University of Maryland post-transplant clinic.

SUMMARY:
Intra-patient variability (IPV) in tacrolimus is associated with premature graft loss. The rate of acute rejection episodes is higher in these patients, and acute rejection impacts negatively on graft survival. The prevalence of patients with high IPV is higher in African American patients (1-5). At the kidney transplant program of the University of Maryland, our investigators follow over 2.800 patients, with approximately 50% of the patients being of African American heritage, thus an ideal setting for the study.

DETAILED DESCRIPTION:
Study Population: Kidney transplant recipients with stable renal function with regular follow-up at the University of Maryland post-transplant clinic with at least 3 levels deemed as appropriately 12-hour trough levels within 3-36 months post-transplant.

Group 1 - patients with high IPV (designated as ≥ 30%). Group 2 - patients with normal IPV (< 30%). Will assess risk of subclinical acute rejection in patients with high IPV compared to normal IPV. All tacrolimus 12 h trough levels in patients with stable allograft function at least 3 months post-transplant.

Calculation of IPV: CV (%) = (SD/mean Tac trough concentration) x 100 (if stable total daily dose). To take into account dose changes, obtained levels will be corrected for the corresponding daily dose of tacrolimus to help correctly calculate IPV (CV C0/D-IPV) (6-7).

Patients will be tested with TruGraf one time during the study.

ELIGIBILITY:
Inclusion Criteria: Patients who meet all of the following criteria are eligible for enrollment:

1. Are males or females of at least 18 years of age.
2. Have the ability to understand the requirements of the study and are able to provide written informed consent.
3. Recipient of a primary or subsequent deceased-donor or living donor kidney transplantation.
4. Stable serum creatinine (current serum creatinine <2.3 mg/dl, <20% increase compared to the average of the previous 3 serum creatinine levels)
5. Kidney transplant patients who >90 days (+/- 2 weeks) post-transplant will be included in this study
6. Patients with at least 3 tacrolimus trough levels( deemed as appropriately 12-hour trough levels) within 3-36 months post-transplant

Exclusion Criteria: Patients who meet any of these criteria are not eligible for enrollment:

1. Inability or unwillingness to provide informed consent.
2. Need for combined organ transplantation with an extra-renal organ and/or islet cell transplant.
3. Recipients of previous non-renal solid organ and/or islet cell transplantation.
4. Infection with HIV.
5. Infection with BK nephropathy.
6. Patients that have nephrotic range proteinuria (urine protein >3 gm/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
TruGraf test validity on immunosuppression damage | up to 18 months post-transplant
  The TruGraf test is a non-invasive blood test that measures molecular gene expression profiles associated with clinical conditions previously only diagnosed by biopsy in kidney transplant recipients. The results of the TruGraf test provide additional information about the adequacy of immunosuppression and may be used to support decisions in patient management.

SECONDARY OUTCOMES:
Renal function associated with premature graft loss | up to 18 months post-transplant
  Utilization of TruGraf testing in patients with stable creatinine, high and normal intrapatient variability (IPV) in tacrolimus levels, between 3 and 18 months post-transplant. This information will aid in determining if local practices should be updated for patient care

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No